CLINICAL TRIAL: NCT06457698
Title: Temporomandibular Bioviscosuplementation (Platelet-Rich Plasma Combined With Hyaluronic Acid) After Double-Puncture Arthrocentesis: a Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Portugues da Face (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUPERPRP
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Hyaluronic acid; platelet-rich plasma; arthrocentesis; viscosuplementation
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects were randomly assigned into two groups: HA injection or HA injection + PRP. Codes were prepared and distributed in the two groups for this allocation. The treatment assignment was made by an independent person who was not involved in performing any other procedures in the study, such as the preoperative injection or the TMJ arthrocentesis. An envelope containing a code was selected and assigned to the patient. Subjects were blinded until the end of the study. The surgeon was unblinded because they could distinguish the color of the two viscosupplements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA injection (Placebo Comparator): After TMJ double-puncture arthrocenthesis under local anesthesia, hyaluronic acid (Suplasyn®, 20 mg/ml) will be injected in the joint with the first portal.
  Interventions: Procedure: Double-puncture TMJ arthrocentesis under local anaesthesia
- HA + PRP injection (Active Comparator): 32ml of venous blood per joint will be collected and added to four 8ml-collection tubes containing sodium citrate. Then, blood will be centrifugated at 800rpm for 8 minutes at room temperature. 3 layers are perceptible: (1)layer with platelet-rich plasma and growth factors; (2)layer with white blood cells; (3)layer corresponding to red blood cells. Then, the total plasma volume will be calculated, and the plasma corresponding to the first fraction (low platelet fraction) aspirated. The second fraction of the first layer corresponding to PRP, above the white blood cell layer, will be removed and transferred to new tubes.
  10 minutes before the mixing with HA, a calcium chloride-rich activator (Endoret ®, BTI Biotechnology Institute, Vitoria-Gasteiz, Álava, Spain) will be added to the PRP. The mixture of PRP with HA was then carried out at a ratio of 1cc of low molecular weight HA (Suplasyn®, 20 mg/ml) +1cc of PRP and introduced in the joint with the first portal.
  Interventions: Procedure: Double-puncture TMJ arthrocentesis under local anaesthesia

INTERVENTIONS:
Procedure: Double-puncture TMJ arthrocentesis under local anaesthesia — The first puncture involved carefully palpating the lateral rim of the glenoid fossa. A 5-cc syringe was prepared with a mixture of 3 cc of Ringer lactate and 1.8 cc of lidocaine with epinephrine. A 21-G needle connected to the syringe was gently inserted into the TMJ skin area. Once the needle tip made contact with the posterior slope of the eminence of the upper joint compartment, it was oriented vertically to access the upper compartment, allowing the surgeon to perform a validation step. For the second puncture, the joint was maintained at maximum distention with continuous inflow through the first portal, while the surgeon felt insufflation/distention in the anterior joint area. The second portal was established using a 21-G needle with successful fluid outflow. After completing an effective circuit, joint washing was carried out using intra-articular hydraulic pressure with at least 150 ml of Ringer lactate solution.

SUMMARY:
Intra-articular injections of hyaluronic acid (HA) or platelet-rich plasma (PRP) have been used with temporomandibular joint (TMJ) arthrocentesis to improve lubricative properties and influence regenerative processes. A randomized, controlled clinical trial investigated the benefits of complementary bioviscosuplementation (HA+PRP) in patients submitted to double-portal TMJ arthrocentesis.

ELIGIBILITY:
Inclusion Criteria:

* (1) age >18 years; (2) history of conservative treatment for TMD without significant improvement for at least three months; (3) clinical diagnosis of unilateral or bilateral intra-articular disorder; (3) clinical criteria for unilateral or bilateral TMJ arthrocentesis; (4) magnetic resonance imaging (MRI) and computed tomography (CT) documenting arthrogenous derangement.

Exclusion Criteria:

* The exclusion criteria included: 1) any history of previous TMJ surgical intervention or any facial trauma within the last 4 weeks before the study; 2) concomitant other contralateral TMJ surgery; 3) severe medical problems or mental illness and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
TMJ arthralgia (VAS, 0-10) | TMJ arthralgia will be assessed preoperatively (T0) and postoperatively (T1 - 1 month, T2 - 3 months, T3 - 6 months, T4 - 12 months follow-up).
  The level of TMJ arthralgia was registered through pain during palpation of the lateral pole or around the lateral pole or pain on maximum unassisted or assisted opening, right or left lateral movements, or protrusive movements, following the DC/TMD guidelines.12, 13 Patient scored for each side using a 10-point VAS, from 0-no pain and 10-severe pain.

SECONDARY OUTCOMES:
maximum mouth opening (MMO) | MMO will be assessed preoperatively (T0) and postoperatively (T1 - 1 month, T2 - 3 months, T3 - 6 months, T4 - 12 months follow-up).
  MMO was measured using a certified ruler between the incisor's teeth.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Português da Face, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No